CLINICAL TRIAL: NCT06570200
Title: Evaluation of Injectable PRF With Vitamin D As an Adjunct to Non-Surgical Therapy in the Treatment of Stage III Periodontitis. A Randomized Controlled Clinical Trial
Brief Title: Evaluation of iPRF With Vit.D As an Adjunct to Non-Surgical Therapy in the Treatment of Stage III Periodontitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed hamed fattouh hamed, dentist, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CairoU50022
Record Dates: First submitted 2024-08-15; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Pocket
Keywords: iPRF; vitamin D; Cholecalciferol; periodontal pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the masking will be applied in the two test groups where iPRF will be used and neither the principle investigator nor the participants will know if vitamin D will be applied to the iPrf or a placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PMPR only (Active Comparator): scaling and root planing only will be made for group 1 (control group)
  Interventions: Procedure: PMPR only
- PMPR + iPRF (Experimental): scaling and root planing plus locally applied iPRF in the periodontal pocket will be made for test group 1.
  Interventions: Procedure: PMPR+iPRF
- PMPR + iPRF + Vit.D (Experimental): scaling and root planing plus locally applied iPRF and vitamin D in the periodontal pocket will be made for test group 2.
  vitamin D will be obtained from a commercial product in the Egyptian pharmacies called (Devarol S) in the form of injectable ampoules containing 200000 IU of cholecalciferol (2.5 mg/ml)
  Interventions: Drug: PMPR+iPRF+Vit.D

INTERVENTIONS:
Procedure: PMPR+iPRF — locally applied iPRF in the periodontal pocket
  Other Names: scaling plus locally applied iPRF
  Arms: PMPR + iPRF
Drug: PMPR+iPRF+Vit.D — locally applied iPRF plus vitamin D in the periodontal pocket
  Other Names: scaling plus locally applied iPRF nd vitamin D
  Arms: PMPR + iPRF + Vit.D
Procedure: PMPR only — scaling and root planing only will be done for the periodontal pocket for the control group
  Other Names: scaling only
  Arms: PMPR only

SUMMARY:
a clinical trial will be made to investigate the effect of locally applied injectable prf (iPRF) plus vitamin D on the periodontal pockets in stage III periodontitis patients

DETAILED DESCRIPTION:
in this clinical trial, the treatment of periodontal pockets in stage III periodontitis patients will be evaluated. the study participants will be divided in 3 groups:

First group >> will be treated with professional mechanical plaque removal (PMPR) only.

second group >> will be treated with PMPR + locally applied iPRF.

Third group >> will be treated with PMPR + locally applied iPRF + vitamin D.

Then the results will be compared after 6 months of the treatment (clinically and radiographically).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy systemic condition.
2. Adult patients ˃ 18 years old.
3. Patients with Stage III periodontitis.
4. Patients accept 3-month follow-up period (cooperative patients).
5. Patients provide an informed consent.

Exclusion Criteria:

1. Presence of prosthetic crowns.
2. Extensive interproximal restorations.
3. Periodontal therapy within the last 12 months.
4. Having undergone surgical periodontal therapy or undergoing orthodontic treatment.
5. Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis.
6. The use of antibiotics or anti-inflammatory drugs 3-month prior to the procedure and till the end of 6-month of follow-up.
7. Smokers.
8. Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
pocket depth reduction | 6 months
  estimate the amount of reduction of the pocket depth from baseline and after 6 months of treatment

SECONDARY OUTCOMES:
clinical attachment level (CAL) gain | 6 months
  the amount of CAL gained from baseline and after 6 months of treatment
Plaque index | 6 months
  comparison of amount of plaque before and after treatment using plaque score
Bleeding on probing (BOP) | 6 months
  measuring the percentage of BOP using a periodontal probe before and after treatment
Gingival Marginal Level (GML) | 6 months
  determining the location of gingival margin in relation to the tooth before and after treatment
Post-operative Pain | 6 months
  comparing the pain before and after treatment using Visual Analogue Scale(VAS) Questionnaire. A scale from 0-10 will be used with 0 means no pain and 10 means maximum pain.
Treatment time taken for each groups | 6 months
  a timer will be used to determine the required time of each procedure of the 3 study groups
degree of bone fill or loss | 6 months
  using digital software, evaluation of the radiographic changes will be done at the area diagnosed with periodontal problem and selected for the treatment before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr Manal Hosny, professor, Study Director — Cairo University; Prof.Dr Karim Fawzy, Professor, Study Director — Cairo University; Prof.Dr Luigi Nibali, Professor, Study Director — King's College London; Dr.Manar T El-zanaty, Doctorate, Study Director — Cairo University; Ahmed Fattouh, Bachelor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torumtay Cin G, Lektemur Alpan A, Cevik O. Efficacy of injectable platelet-rich fibrin on clinical and biochemical parameters in non-surgical periodontal treatment: a split-mouth randomized controlled trial. Clin Oral Investig. 2023 Dec 28;28(1):46. doi: 10.1007/s00784-023-05447-8. PMID 38153510